CLINICAL TRIAL: NCT04442321
Title: Effectiveness of Ultrasound-Guided Percutaneous Electrical Stimulation on Radial Nerve With Exercises in Patients With Lateral Epicondylalgia
Brief Title: Ultrasound-Guided Percutaneous Electrical Stimulation on Radial Nerve in Patients With Lateral Epicondylalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 19/043
Record Dates: First submitted 2020-05-21; First posted 2020-06-22 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2023-12

CONDITIONS: Tennis Elbow
Keywords: Lateral Epicondylalgia; Lateral Epicondylitis; Lateral Elbow Tendinopathy; Lateral Elbow Pain; Percutaneous Electrical Nerve Stimulation
MeSH Terms: conditions — Tennis Elbow | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PENS plus exercise group (Active Comparator): Experimental: PENS plus exercise group 4-week intervention program with 1 weekly treatment session, one of percutaneous electrical stimulation. In addition, self-management loaded exercise, prescribed by the physical therapist but completed by the patient independently . It involved isometric exercises, eccentric exercise, eccentric-concentric with weight or resistive therapeutic band.
  Interventions: Other: PENS plus exercise
- Sham PENS plus exercise group (Sham Comparator): Sham Comparator: Sham PENS plus exercise group 4-week intervention program with 1 weekly treatment session, one of percutaneous electrical stimulation. In addition, self-management loaded exercise, prescribed by the physical therapist but completed by the patient independently. It involved isometric exercises, eccentric exercise, eccentric-concentric with weight or resistive therapeutic band.
  Interventions: Other: Sham PENS plus exercise

INTERVENTIONS:
Other: PENS plus exercise — The technique will be performed ultrasound-guided on the radial nerve, the places of the needle's insertions will be the following:
  * Needle will be placed at under the lateral intermuscular septum between the triceps brachii and brachialis, approximately 10cm superior to the lateral epicondyle
  * Needle will be placed at the upper third of the forearm on the posterior interosseous nerve after passing the arcade of Froshe
  The percutaneous electrical stimulation will be realized with a transcutaneous electric nerve stimulation (TENS) current:
  * TENS Frequency 2 Hz
  * TENS Pulse width - 250 microseconds
  * Duration - 30 minutes.
  * TENS Intensity - Increased at an intensity of visible motor response of the innervated musculature and maximal tolerable intensity.
  * Administration - One per week
  Self-management loaded exercises prescribed by a physical therapist, two times per week.
  Arms: PENS plus exercise group
Other: Sham PENS plus exercise — The technique will be performed ultrasound-guided on the radial nerve, the places of the needle's insertions will be the following:
  * Needle will be placed at under the lateral intermuscular septum between the triceps brachii and brachialis, approximately 10cm superior to the lateral epicondyle
  * Needle will be placed at the upper third of the forearm on the posterior interosseous nerve after passing the arcade of Froshe
  The electrical current will not be working, and the needles will be placed during 30 minutes:
  - Administration - One per week
  Self-management loaded exercises prescribed by a physical therapist, two times per week.
  Arms: Sham PENS plus exercise group

SUMMARY:
Lateral epicondylalgia is a common musculoskeletal condition that approximately affects 1-3% of the general population. Several authors have found greater mechanical pain sensitivity in the radial nerve when compared with healthy subjects. Radial tunnel syndrome exhibits a similar clinical presentation to lateral epicondylalgia. Percutaneous electrical stimulation has shown reduce pain in several conditions. Percutaneous electrical stimulation on the radial nerve could cause an important relief in lateral epicondylalgia.

Hypothesis: Percutaneous electrical stimulation on radial nerve plus exercise therapy in patients with lateral epicondylalgia is better than sham percutaneous electrical stimulation plus exercise.

DETAILED DESCRIPTION:
Randomized, double-blind, placebo controlled clinical trial, using Percutaneous Electrical Nerve Stimulation (PENS). PENS is technique to provide a transcutaneous electrical nerve stimulation current throughout needling filaments place close to the nerve.

Study Aims:

Aim #1: The primary aim of the study is to compare the effect of the short, mid and long-term of PENS on intensity of pain as measured by numeric pain rating scale and disability as measured by Patient Rated Tennis Elbow Evaluation (PRTEE) in patients with lateral epicondylalgia with random assignment to two treatments: PENS plus exercise program or Sham PENS plus exercise program.

Aim #2: The secondary aim of the study is to compare the effect of the short, medium and long-term of PENS on disability as measured by DASH questionnaire, and psychological factors (fear and avoidance and catastrophism) and Global Rating of Change (GRoC) in patients with lateral epicondylalgia with random assignment to two treatments: PENS plus exercise program or Sham PENS plus exercise program.

ELIGIBILITY:
Inclusion Criteria:

* Lateral epicondylalgia symptoms confirmed with at least 2 of the 4 following test:

  1. pain during palpation of lateral epicondyle
  2. pain on resisted wrist extension
  3. pain on resisted middle finger extension
  4. pain during hand-grip.

Exclusion Criteria:

* History of fractures, luxations, surgery and/or musculoskeletal disorders in upper limb.

  * Neurological disorders, inflammatory and/or degenerative diseases.
  * Having received as treatment techniques that involve needles on the previous 6 months to study enrollment, or having received percutaneous electrical stimulation as a treatment before.
  * Cervical pathology, fibromyalgia, unstable cardiovascular diseases, pregnant women or under suspect of pregnancy.
  * Contraindications of needle's insertions: anticoagulant therapy, needle phobia, diabetes, hypothyroidism, lymphoedema, muscular diseases).
  * Contraindications of electrical current application.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Changes in Elbow Pain Intensity between baseline and follow-up periods | Baseline, 1 week post-intervention, and 1, 3, 6 and 12 months after the intervention
  Pain intensity measured with a 10 (0 - No pain - 10 The worst pain) numeric rating scale

SECONDARY OUTCOMES:
Changes in Elbow Related-Disability between baseline and follow-up periods | Baseline,1 week post-intervention, and 1, 3, 6 and 12 months after the intervention
  Measured with Patient Rated Tennis Elbow Evaluation (PRTEE). It is a 15-item questionnaire designed to measure forearm pain and disability in patients
Changes in Upper Extremity Related-Disability between baseline and follow-up period | Baseline, 1 week post-intervention, and 1, 3, 6 and 12 months after the intervention
  Measured with Disabilities of the Arm, Shoulder and Hand (DASH) Questionnaire. It includes 30 items assessing (1) degree of difficulty during the preceding week in performing several physical activities because of problems in a upper extremity (21 items), (2) severity of each of the symptoms of pain, activity related pain, tingling, weakness, and stiffness (5 items), and (3) the problem's effect on social activities, work, and sleep and its psychological impact (4 items). Each item is answered on a 5-point scale ranging from 1 (no difficulty to perform, no symptom, or no impact) to 5 (unable to do, very severe symptom, or high impact). The responses to the 30 items are summed to form a raw score that is then converted to a scale from 0 to 100 with a formula. A higher score reflects greater disability.
Changes in Kinesiophobia between baseline and follow-up periods | Baseline,1 week post-intervention, and 1, 3, 6 and 12 months after the intervention
  Tampa Scale for Kinesiophobia. To assess the fear of movement and pain-related fear. The 11 items are scored 1-4, with total scores ranging from 11 to 44. The addition of all the points obtained from each of the items results in the level of kinesiophobia, with higher scores indicating greater perceived kinesiophobia
Changes in Pain Catastrophizing between baseline and follow-up periods | Baseline, 1 week post-intervention, and 1, 3, 6 and 12 months after the intervention
  Pain Catastrophizing Scale (PCS). This tool is a 13-item questionnaire designed to measure the three components of pain-related catastrophizing: rumination, magnification, and helplessness, resulting in a unique score. Each item is responded to on a 5-point scale (0 not at all, 4 all the time) relating the degree to which the individual experiences a thought or feeling of a painful situation.
Changes in Self-perceived Improvement between baseline and follow-up periods | Baseline,1 week post-intervention, and 1, 3, 6 and 12 months after the intervention
  Global ratings on changes in regards to their level of elbow well-being since the treatment on a 15-point self-report scale (from -7, very much worse, to 7, completely recover)

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Complutense de Madrid, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No